CLINICAL TRIAL: NCT04437056
Title: Outcome Measurements After Cognitive Nerve Transfers to Spastic Muscles in Stroke Patients
Brief Title: Nerve Transfers in Post-stroke Spasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Vienna (Other)
Collaborators: Imperial College London (Other); Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Olga Politikou, MD, Principal Investigator, PhD Student Clinical Laboratory for Bionic Extremity Reconstruction, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK 2319/2019
Record Dates: First submitted 2020-06-01; First posted 2020-06-18 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Spasticity as Sequela of Stroke; Nerve Transfers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke patients with upper limb spasticity (Other): Patients with post-stroke upper limb spasticity will be operated for cognitive nerve transfers to spastic muscles to allow for volitional muscle reinnervation and disrupture of spasticity. Adequate healthy nerve donors from the ipsilateral arm will be determined clinically and electrophysiologically.
  Interventions: Procedure: Cognitive nerve transfers to spastic upper extremity muscles in stroke patients

INTERVENTIONS:
Procedure: Cognitive nerve transfers to spastic upper extremity muscles in stroke patients — Based on the fact that upper motor neuron syndrome after stroke is presented with variable clinical features, usually without affecting in the same way the entire upper extremity, we aim to investigate the efficacy of nerve transfers to spastic muscles after stroke using as donor nerves that innervate unaffected ipsilateral volitionally controlled muscles.

SUMMARY:
Stroke is nowadays a leading cause of disability with devastating sequelae. Upper limb spasticity is one of them. Nevertheless, not all the muscles are equally affected, as some may turn spastic or paretic and other remain intact. This unique pathophysiological mosaic dictates a precise therapeutic plan. Existing spasticity treatment has significant drawbacks due to its unspecific targeting and short duration. A causal, life-lasting treatment, precisely adapted to every single patient's needs and to disease pattern, is currently missing. Hyperselective muscle denervation and subsequent cognitive reinnervation with appropriate unaffected donor nerves may break the pathological spastic circuit and provide volitional muscle control. With this pioneering study we will perform cognitive nerve transfers to spastic muscles and will prospectively investigate their effects on clinical, electrophysiological, molecular-biological and histological level. Accurate donor nerve selection will be for the first time quantified through motor unit number estimation with high-density needle electromyography. This revolutionary concept can open the window to a new era of therapeutic possibilities for stroke victims.

ELIGIBILITY:
Inclusion Criteria:

* Are undergoing nerve transfers
* Age from 18 to 75 years old
* Minimum of 1 year interval after stroke
* Are able to understand German or English
* Medical Research Council (MRC) Muscle scale for donor nerves: M4 or M5
* Walking patients, with or without crutches
* Good general health condition and social support

For the control group:

* Age 18-75 years old
* Indication for ulnar nerve release and submuscular transposition for compression neuropathy in the elbow
* No other neurological disorders

Exclusion Criteria:

* Stroke earlier than 3 years at the time of first consultation
* Lower limb spasticity and patients mobile with wheel chair

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Chedoke Arm and Hand Activity Inventory (CAHAI-9) score | 0-24 months
  Patients can reach a score for CAHAI 9 between 9 to 63. The lower the score, the greater impairment.
Modified Ashworth Scale | 0-24 months
  A score of 1 indicates no resistance, and 5 indicates rigidity. A 1+ scoring category indicates resistance through less than half of the movement. Scores range from 0-4, with 6 choices .
Changes in electrophysiological muscle activity after nerve transfers | 0-24 months
  Low frequency-dependent depression of H-wave (in mV)

SECONDARY OUTCOMES:
Changes in muscle satellite cell population (%) in spastic muscles and comparison with healthy control group | During surgery- 24 months
  Muscle biopsies from spastic muscles will be obtained during the surgery of nerve transfers. The muscle satellite cell population (%) will be calculated with the use of Flow Cytometry and be compared to the one of healthy muscles of control group. There will be no recruitment procedure for the control group. Routinely, when we carry out surgery for ulnar nerve release in the elbow and nerve transposition, a part of the flexor carpi ulnaris muscle needs to be excised and discarded. After obtaining informed consent from patients for further use of their biological material, we will collect these muscles and use them as control group.
The Action Research Arm Test (ARAT) | 0-24 months
  The total score on the ARAT ranges from 0 to 57, with the lowest score indicating that no movements can be performed, and the upper score indicating normal performance.
The Disabilities of the Arm, Shoulder and Hand (DASH) score | 0-24 months
  Scores range from 0 (no disability) to 100 (most severe disability).
Motor Unit Number Estimation of donor and spastic muscles | 0-24 months
  High density electromyography with fine needle electrodes will be applied to allow an accurate estimation of motor units (absolute number) in donor muscles, in spastic muscles and in newly-innervated muscles
Comparison of collagen content between spastic and healthy muscles | During surgery- 12 months
  Muscle biopsies from spastic muscles will be obtained during the surgery of nerve transfers. Collagen content of spastic muscles (%) will be calculated with the use of Picrosirius red staining and bright field light microscopy and be compared with healthy muscles of control group. There will be no recruitment procedure for the control group. Routinely, when we carry out surgery for ulnar nerve release in the elbow and nerve transposition, a part of the flexor carpi ulnaris muscle needs to be excised and discarded. After obtaining informed consent from patients for further use of their biological material, we will collect these muscles and use them as control group.
Changes in sarcomere length (μm) in spastic muscles | During surgery- 12 months
  Biopsy of a muscle fascicle from spastic muscles will be obtained during the surgery of nerve transfers with the use of dedicated clamps and will be fixed in formalin. The sarcomere length will be calculated with the use of fractional laser. The sarcomere length of spastic muscles will be compared with the sarcomere length of healthy control group muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Aszmann, Prof, Study Director — Department of Surgery, Medical University of Vienna
Locations (1):
- General Hospital of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urban PP, Wolf T, Uebele M, Marx JJ, Vogt T, Stoeter P, Bauermann T, Weibrich C, Vucurevic GD, Schneider A, Wissel J. Occurence and clinical predictors of spasticity after ischemic stroke. Stroke. 2010 Sep;41(9):2016-20. doi: 10.1161/STROKEAHA.110.581991. Epub 2010 Aug 12. PMID 20705930
- [Background] Wissel J, Manack A, Brainin M. Toward an epidemiology of poststroke spasticity. Neurology. 2013 Jan 15;80(3 Suppl 2):S13-9. doi: 10.1212/WNL.0b013e3182762448. PMID 23319481
- [Background] Sommerfeld DK, Gripenstedt U, Welmer AK. Spasticity after stroke: an overview of prevalence, test instruments, and treatments. Am J Phys Med Rehabil. 2012 Sep;91(9):814-20. doi: 10.1097/PHM.0b013e31825f13a3. PMID 22760104
- [Background] Zheng MX, Hua XY, Feng JT, Li T, Lu YC, Shen YD, Cao XH, Zhao NQ, Lyu JY, Xu JG, Gu YD, Xu WD. Trial of Contralateral Seventh Cervical Nerve Transfer for Spastic Arm Paralysis. N Engl J Med. 2018 Jan 4;378(1):22-34. doi: 10.1056/NEJMoa1615208. Epub 2017 Dec 20. PMID 29262271
- [Background] Qiu YQ, Du MX, Yu BF, Jiang S, Feng JT, Shen YD, Xu WD. Contralateral Lumbar to Sacral Nerve Rerouting for Hemiplegic Patients After Stroke: A Clinical Pilot Study. World Neurosurg. 2019 Jan;121:12-18. doi: 10.1016/j.wneu.2018.09.118. Epub 2018 Sep 26. PMID 30266703
- [Background] Khalifeh JM, Dibble CF, Van Voorhis A, Doering M, Boyer MI, Mahan MA, Wilson TJ, Midha R, Yang LJS, Ray WZ. Nerve transfers in the upper extremity following cervical spinal cord injury. Part 1: Systematic review of the literature. J Neurosurg Spine. 2019 Jul 12;31(5):629-640. doi: 10.3171/2019.4.SPINE19173. Print 2019 Nov 1. PMID 31299644
- [Background] Faturi FM, Lopes Santos G, Ocamoto GN, Russo TL. Structural muscular adaptations in upper limb after stroke: a systematic review. Top Stroke Rehabil. 2019 Jan;26(1):73-79. doi: 10.1080/10749357.2018.1517511. Epub 2018 Sep 17. PMID 30222075
- [Background] Smith LR, Pichika R, Meza RC, Gillies AR, Baliki MN, Chambers HG, Lieber RL. Contribution of extracellular matrix components to the stiffness of skeletal muscle contractures in patients with cerebral palsy. Connect Tissue Res. 2021 May;62(3):287-298. doi: 10.1080/03008207.2019.1694011. Epub 2019 Nov 28. PMID 31779492
- [Background] Mandeville RM, Brown JM, Sheean GL. Semi-quantitative electromyography as a predictor of nerve transfer outcome. Clin Neurophysiol. 2019 May;130(5):701-706. doi: 10.1016/j.clinph.2019.02.008. Epub 2019 Feb 28. PMID 30875537
- [Background] Barreca S, Gowland CK, Stratford P, Huijbregts M, Griffiths J, Torresin W, Dunkley M, Miller P, Masters L. Development of the Chedoke Arm and Hand Activity Inventory: theoretical constructs, item generation, and selection. Top Stroke Rehabil. 2004 Fall;11(4):31-42. doi: 10.1310/JU8P-UVK6-68VW-CF3W. PMID 15592988